CLINICAL TRIAL: NCT01717872
Title: Comparing the Laryngoscopy View Using Miller and Macintosh Laryngoscopy Blades in Infants Under Two Years of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jerrold Lerman, Clinical Professor of Anesthesiology, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lerman Blade study
Record Dates: First submitted 2012-10-28; First posted 2012-10-31 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Percent of Glottic Opening
Keywords: glottis, laryngoscopy, laryngoscope blade

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Macintosh laryngoscope blade (Active Comparator): A photo of the larynx will be taken with the Macintosh laryngoscope blade lifting and not lifting the epiglottis. The view of the larynx will be assessed using the Percent of Glottic Opening (POGO) score by a blinded assessor.
  Interventions: Device: Laryngoscope blade
- Miller laryngoscope blade (Active Comparator): A photo of the larynx will be taken with the Miller laryngoscope blade lifting and not lifting the epiglottis. The view of the larynx will be assessed using the percent of glottic opening score by a blinded assessor.
  Interventions: Device: Laryngoscope blade

INTERVENTIONS:
Device: Laryngoscope blade — The POGO score will be used to assess the percent of the glottis that can be seen with each of the blades lifting and not lifting the epiglotis
  Other Names: Macintosh laryngoscope blade; Miller laryngoscope blade

SUMMARY:
To compare the laryngoscopy view using two standard clinical devices, the Macintosh and Miller laryngoscopy blades, in infants between one day and two years of age.

Miller blades (straight blades) are more commonly used than MacIntosh blades (curved) in pediatric clinical practice in some institutions especially in infants. The anatomy of infant airway has traditionally been considered to lend itself to advantages of the Miller blade. Some argue that the Miller blade offers a superior view of the laryngeal inlet because it lifts the epiglottis. However, others use the Miller blade to expose the larynx without lifting the epiglottis, supposedly to avoid traumatizing it. Despite the long-standing use of these blades, more than 50 years, no systematic study has ever compared the laryngoscopy views of the Miller and Macintosh blades in infants.

DETAILED DESCRIPTION:
* After Institutional Review Board approval, the patients meeting inclusion criteria will be selected from the Operating room elective surgical list.
* They will be randomized to one of the two groups: a #1 Miller or Macintosh blade.
* After obtaining informed consent from the parent or the legal guardian, monitors (electrocardiogram, non-invasive blood pressure monitor and pulse oximeter) that are routine induction of anesthesia will be applied and anesthesia will be induced using an inhalation technique with sevoflurane, nitrous oxide and oxygen. An intravenous cannula will then be placed. The child will then receive a standard intubating dose of a muscle relaxant (rocuronium 0.5-1 mg/kg). The lungs will be mask ventilated using 100% oxygen in Sevoflurane for 3 minutes to allow appropriate time for the muscle relaxant to be fully effective. At that time, the randomized code for that child will be opened and laryngoscopy will be performed with either a Miller or MacIntosh blade as indicated by the code.
* The best possible glottic view will be obtained by ensuring the following steps. The child's head will be positioned in the Magill position, muscle relaxant will be administered, firm forward traction will be applied to the laryngoscope handle, and if needed, external laryngeal manipulation will be applied.
* During the same laryngoscopy, the best glottic visualization will be obtained with the blade lifting the epiglottis and not lifting the epiglottis, in random order (by flipping a coin). This difference is a matter of moving the position of the blade back without removing the blade from the larynx.
* The two views will be recorded by a second doctor using a SONY camera at the mouth adjacent to the laryngoscope handle.
* Photos of the glottic opening will be graded using the POGO scale (Ref1) by a third (blinded) anesthesiologist.
* All of the intubations and image acquisition will be performed by Drs. Yuvesh Passi, Jerrold Lerman or Chris Heard.
* The images obtained will not have patient identifiers included. They will be stored in a secure file once the study is completed that will be accessed only by investigators involved in the study.
* No patient identifiers will be included on any documentation apart from the source documents.
* The research data will be stored in a locked office of Dr. Lerman (Room 251) in Department of Anesthesia, Women and Children's Hospital of Buffalo during and after the study for security to protect subject privacy and confidentiality.
* There will be no payments or compensation to the study subjects

The primary hypothesis of this study is to compare the view of the larynx with Miller blade while lifting the epiglottis to the Macintosh blade lifting the tongue, in infants and children <2 years of age. However, views will be obtained with the Miller and Macintosh blades both lifting and not lifting the epiglottis and comparisons between pairs of measurements will be performed. In order for to detect superiority of one technique over the other, we will need a difference in the POGO scores of 25 points with a standard deviation of 25 points, yielding a sample size of 15 children in each group. To account for photographic difficulties, unreadable photos as well as dropouts, we will enroll 25 children in each group. Therefore a total of 50 children will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists physical status 1 and 2 infants and children
* Age <2 years of age
* All racial and ethnic origin
* Scheduled for elective surgery
* Fasting patients who are unmedicated preoperatively

Exclusion Criteria:

* History of difficult airway
* Severe asthma
* Premature birth
* ICU stay for more than a week following delivery
* Acute or chronic pulmonary or neuromuscular diseases

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Lerman, MD, Principal Investigator — SUNY at Buffalo, Women and Children's Hospital of Buffalo
Locations (1):
- Women and Childrens Hospital of Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Passi Y, Sathyamoorthy M, Lerman J, Heard C, Marino M. Comparison of the laryngoscopy views with the size 1 Miller and Macintosh laryngoscope blades lifting the epiglottis or the base of the tongue in infants and children <2 yr of age. Br J Anaesth. 2014 Nov;113(5):869-74. doi: 10.1093/bja/aeu228. Epub 2014 Jul 25. PMID 25062740

RESULTS

PARTICIPANT FLOW:
Groups:
- Macintosh Laryngoscope Blade: A photo of the larynx will be taken with the Macintosh laryngoscope blade lifting and not lifting the epiglottis. The view of the larynx will be assessed using the POGO score by a blinded assessor.
  Laryngoscope blade: The POGO score will be used to assess the percent of the glottis that can be seen with each of the blades while lifting or not lifting the epiglottis
- Miller Laryngoscope Blade: A photo of the larynx will be taken with the Miller laryngoscope blade lifting and not lifting the epiglottis. The view of the larynx will be assessed using the POGO score by a blinded assessor.
  Laryngoscope blade: The POGO score will be used to assess the percent of the glottis that can be seen with each of the blades while lifting or not lifting the epiglottis
Period: Overall Study
Arm/Group | Macintosh Laryngoscope Blade | Miller Laryngoscope Blade
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Macintosh Laryngoscope Blade | Miller Laryngoscope Blade | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Full Range); unit: months]
  Age | 15 [4 to 23] | 14 [5 to 23] | 14 [4 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 16 | 19 | 35
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
percent of glottic opening [Median (Inter-Quartile Range); unit: percentage] | 80 [80 to 100] | 80 [60 to 100] | 80 [60 to 100]

OUTCOME MEASURES:

1. Primary Outcome: The View of the Larynx (Glottis Opening) as Determined by POGO Score (Percentage of Glottic Opening).
Description: Percent of glottic opening (POGO) with the Miller blade lifting the epiglottis compared with the score with the Macintosh blade lifting the tongue
Time Frame: 30 seconds
Measure: Mean (95% Confidence Interval); unit: percentage of Glottic opening
Groups:
- Macintosh Laryngoscope Blade: A photo of the larynx will be taken with the Macintosh laryngoscope blade lifting and not lifting the epiglottis. The view of the larynx will be assessed using the POGO score by a blinded assessor.
  Laryngoscope blade: The percent of glottic opening (POGO) score will be used to assess the percent of the glottis that can be seen with each of the blades while lifting or not lifting the epiglottis
Arm/Group | Macintosh Laryngoscope Blade | Miller Laryngoscope Blade
Number analyzed (Participants) | 25 | 25
percentage of Glottic opening | 84 [76 to 92] | 78 [70 to 87]
Statistical Analysis 1: Comparison: Macintosh Laryngoscope Blade vs Miller Laryngoscope Blade; MAC blade lifting the tongue versus Miller blade lifting the epiglottis; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percent of Glottic Opening With the Miller Blade Lifting the Epiglottis and Tongue
Description: Percent of glottic opening (POGO) with the Miller blade lifting the epiglottis compared with the score with the same blade lifting the tongue
Time Frame: 30 seconds
Measure: Mean (95% Confidence Interval); unit: percent of glottic opening
Groups:
- Miller Blade Lifting the Epiglottis: Miller blade was inserted under the epiglottis to lift it to view the glottic opening
- Miller Blade Lifting the Tongue: Miller blade was inserted under the tongue (above the epiglottis) to view the glottic opening
Arm/Group | Miller Blade Lifting the Epiglottis | Miller Blade Lifting the Tongue
Number analyzed (Participants) | 25 | 25
percent of glottic opening | 78.4 [70 to 87] | 76 [67.1 to 84.9]
Statistical Analysis 1: Comparison: Miller Blade Lifting the Epiglottis vs Miller Blade Lifting the Tongue; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percent of Glottic Opening With the MAC Blade Lifting the Tongue and the Epiglottis
Description: The MAC blade was inserted under the tongue to view the percent glottic opening and compared with the view with the same blade lifting the epiglottis to view the percent glottic opening.
Time Frame: 30 seconds
Measure: Mean (95% Confidence Interval); unit: percent of glottic opening
Groups:
- MAC Blade Lifting the Tongue: The MAC blade was inserted under the tongue and lifted to view the percent glottic opening
- MAC Blade Lifting the Epiglottis: The MAC blade was inserted under the epiglottis and lift to view the percent glottic opening
Arm/Group | MAC Blade Lifting the Tongue | MAC Blade Lifting the Epiglottis
Number analyzed (Participants) | 25 | 25
percent of glottic opening | 84.4 [76.5 to 92.3] | 67.2 [56.1 to 78.3]
Statistical Analysis 1: Comparison: MAC Blade Lifting the Tongue vs MAC Blade Lifting the Epiglottis; Test type: Superiority or Other; p < 0.0004, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Single assessment, immediately after induction of general anesthesia
Arm/Group | Macintosh Laryngoscope Blade | Miller Laryngoscope Blade
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macintosh Laryngoscope Blade (N=25) | Miller Laryngoscope Blade (N=25)
(Respiratory, thoracic and mediastinal disorders) | 0 | 0
(Respiratory, thoracic and mediastinal disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No